CLINICAL TRIAL: NCT06794177
Title: Investigation of the Effects of Dual Task Training With Different Task Priorities on Physical Performance and Cognitive Status in Patients With Parkinson's Disease
Brief Title: The Effects of Dual Task Training With Different Task Priorities on Physical Performance and Cognitive Status in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Gazi University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elvan ÖZCAN GÜLŞEN, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 285
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease (PD); Dual-task; Balance; Walking; Mobility; Cognition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Contol Group (Active Comparator): Single task training
  Interventions: Other: Single task training
- Variable priority dual task training group (Experimental): Variable priority dual task training
  Interventions: Other: Variable priority dual task training
- Fixed priority dual task training group (Experimental): Fixed priority dual task training
  Interventions: Other: Fixed priority dual task training

INTERVENTIONS:
Other: Variable priority dual task training — Variable priority dual task training with balance and walking exercises performed simultaneously with cognitive tasks, twice a week for six weeks
  Arms: Variable priority dual task training group
Other: Fixed priority dual task training — Fixed priority dual task training with balance and walking exercises performed simultaneously with cognitive tasks, twice a week for six weeks
  Arms: Fixed priority dual task training group
Other: Single task training — Single task training with balance and walking exercises, twice a week for six weeks
  Arms: Contol Group

SUMMARY:
This study was planned to investigate and compare the effects of variable and fixed priority dual task training on balance, walking skills, mobility and cognition in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Having agreed to participate in the research after being given detailed information about the research.
* Having been diagnosed with Parkinson's disease by a specialist neurologist according to the UK Brain Bank criteria
* Being in stage 1-3 according to Hoehn & Yahr
* Being 40 years of age or older

Exclusion Criteria:

* Having a neurological condition other than Parkinson's disease
* Cognitive impairment
* Have undergone deep brain stimulation surgery
* Having a visual, auditory or perceptual problem
* Having any orthopedic, rheumatological or other disease that may affect walking and balance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Hoehn and Yahr Scale | Baseline, 6 weeks
  A staging system that quickly provides information in determining the degree and symptom severity of the disease
Unified Parkinson's Disease Rating Scale | Baseline, 6 weeks
  Evaluates cognitive skills, mood, activities of daily living, motor skills, motor fluctuations, dyskinesias, and autonomic dysfunction in four parts
Berg Balance Scale | Baseline, 6 weeks
  It includes 14 functional activities to assess static and proactive balance. The total score ranges from 0 to 56, with higher scores indicating better balance.
Functional Reach Test | Baseline, 6 weeks
  The test is designed to assess dynamic balance by measuring the maximum distance that a person can reach forward beyond arm's length without taking a step.
Single Leg Stance Test | Baseline, 6 weeks
  It is a test method used to evaluate static balance. One foot is lifted without touching the supporting leg and the person is expected to maintain their balance for 30 seconds.
Four Square Step Test | Baseline, 6 weeks
  It is a test method used to evaluate dynamic balance. Two canes are placed on a flat surface to create 4 squares. All squares are numbered. The subject starts in one square and steps in one direction into each of the four squares and then reverses direction back to the start. The time (in seconds) taken to complete the sequence is measured.
10 Meter Walk Test | Baseline, 6 weeks
  Used to assess walking speed. Participants are asked to walk a distance of 10 meters and the time taken is recorded.
Figure-of-Eight Walk Test | Baseline, 6 weeks
  The participant stands still at the midpoint of two cones placed 1.52 m apart and begins walking around the cones in a figure eight at his/her usual pace. The total time and number of steps taken to complete the test are recorded.
3-Meter Backward Walk Test | Baseline, 6 weeks
  The 3-meter distance is measured and marked. Participants are asked to walk backwards as quickly as possible with the "walk" command and to stop when they reach 3 meters. The elapsed time is recorded in seconds.
Timed Up and Go Test | Baseline, 6 weeks
  It is used to assess functional mobility level. The participant is asked to stand up from the chair, walk 3 m, turn around, walk back to the chair and sit down. The test starts with the "walk" command and the completion time is recorded in seconds.
Unified Parkinson's Disease Rating Scale, Part 2 | Baseline, 6 weeks
  UPDRS Part 2 generally is considered a psychometrically reliable tool for measuring activities of daily living outcomes in people with Parkinson's disease.
Dual Task Questionnaire | Baseline, 6 weeks
  It is used to obtain information about the difficulties experienced in daily tasks related to dual task. It consists of 10 questions, each question is scored between 0 and 4.
Trail Making Test | Baseline, 6 weeks
  It is used to evaluate individuals' visual scanning speed, executive functions, visual-motor perception, motor function, planning, organization, abstract thinking and response limitation. The test consists of 2 parts: A and B. In part A, the individual is asked to combine numbers from 1 to 25 and the completion time is recorded. In part B, the individual completes the sequence by corresponding to a number and a letter, and the completion time is recorded.
Stroop Test | Baseline, 6 weeks
  It is a test that evaluates executive functions and the suppression of inappropriate automatic responses and provides information about frontal functions.
Symbol Digit Modalities Test | Baseline, 6 weeks
  It is a test that measures working memory and information processing speed. In the upper right corner of the A4 paper used in the test, there is a grid of shapes, each representing a number. In the other parts of the paper, there are randomly arranged shapes in blocks. During the test, patients are asked to match these shapes with the numbers in the grid.
Word List Generation | Baseline, 6 weeks
  It is a test used to evaluate complex attention functions and vocabulary. It consists of animal and KAS sections. First, the patient is asked to name every animal that comes to mind in one minute, as quickly as possible. In the KAS section, the patient is asked to name every word that comes to mind, except for proper nouns and city names, with the letters K-A-S in order. The time for each letter is again one minute.
Tampa Scale for Kinesiophobia | Baseline, 6 weeks
  It is a 17-question scale developed to measure fear of movement/re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. Each item is scored between 1-4.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Sağlık Bilimleri Üniversitesi, Gülhane Fizyoterapi ve Rehabilitasyon Fakültesi, Ankara
  - Gazi Üniversitesi Tıp Fakültesi Nöroloji Anabilim Dalı, Ankara